CLINICAL TRIAL: NCT05731167
Title: Validation and Application of a Multi-dimentional Frailty Assessment Tool-Cohort Intervention and Follow up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202112187RIND
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Frailty; Fall; Sarcopenia
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular follow up (Active Comparator): Subjects underwent routine outpatient care after assessment and will receive outcomes follow up for 1 year.
  Interventions: Other: Regular follow up
- Multidomain intervention (Experimental): The intervention group will receive multi-faceted frailty prevention programs such as physical training, nutritional advice, cognitive training, and drug education and receive outcomes follow up for 1 year.
  Interventions: Behavioral: Multidomain frailty prevention method

INTERVENTIONS:
Behavioral: Multidomain frailty prevention method — We use the nutrition, physical training, medication consultation, cognition training to prevent the occurrence of frailty or other adverse outcome.
  Arms: Multidomain intervention
Other: Regular follow up — Subjects will receive regular follow up and suggestion in outpatient department.
  Arms: Regular follow up

SUMMARY:
We aim to (1) use a multifaceted, frailty assessment model. (2) use randomized controlled trials to deal with and intervene with cross-field, multi-faceted and intelligent remote management strategies for the elderly with different degrees of frailty, to further observe functional changes and analyze the probability of adverse prognosis such as falls, hospitalization, and death in the future

DETAILED DESCRIPTION:
Background: Frailty is a common problem among the elderly, and it is closely related to their own age, chronic diseases, physical function, and nutritional status. The higher the incidence, the higher the age. Frailty is also associated with many adverse outcomes, such as falls, disability and even mortality. At present, there is no ideal treatment for frailty. It is best to start with prevention and take precautions against various frailty factors in advance. There are two types of frailty assessments in this study. The Clinical Frailty Scale is a single observational assessment method, which can roughly know your frailty degree. Frailty indicators are further combined with questionnaires and instrumental measurements, which can be subdivided to explore different weaknesses such as subjective frailty, objective frailty, sarcopenia, osteoporosis risk, and fall risk for analysis.

Objects: Elderly people in the community (over 65 years old) who seek medical treatment in the Geriatrics Department of National Taiwan University Hospital, and who are willing to accept the frailty index test are eligible for admission. We expect to enroll about 216 cases from 2023.2.1 to 2024.12.31 with intervene and follow up for 1 year.

Method:. All the elders were given questionnaires and instruments to measure various frailty indicators, such as walking speed, standing up and walking test, muscle mass index, grip strength, 5 times of sitting and standing speed, and various physiological indicators such as blood oxygen, body fat, etc. The subjects will be randomly assigned to the intervention group or the control group. The control group will receive routine outpatient care. The intervention group will receive multi-faceted frailty prevention and treatment programs such as physical exercises, nutritional advice, cognitive training, and drug education. After that, the prognosis will be tracked by telephone every 3 months, and the self-evaluation questionnaire and the measurement of frailty indicators will be carried out at the 6th and 12th months. In order to observe the changes in the prognosis and frailty indicators of the two groups in one year.

ELIGIBILITY:
Inclusion Criteria:

* adults aged greater than 65 years in outpatient department

Exclusion Criteria:

* with dementia
* with active cancer and those unable to operate or follow measuring instructions.
* Individuals with pacemakers or metal implants were excluded because those devices may interfere with measurement of body composition using the bioelectrical impedance analysis (BIA) technique

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-02-07 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Fall | 1 year
  fall rate will be evaluated by phone contact to subjects.
Emergency room visits | 1 year
  Emergency room visits will be evaluated by phone contact to subjects.
Hospitalization | 1 year
  Hospitalization times will be evaluated by phone contact to subjects.

SECONDARY OUTCOMES:
Skeletal muscle index | 1 year
  Skeletal muscle index will be measured by Bioelectrical impedance analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Pei Lin, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Kun-Pei Lin, Taipei, Taiwan